CLINICAL TRIAL: NCT04588337
Title: INtravenous TNK for Acute isChemicsTroke in China (INTACT-China): a Prospective, Multi-center, Registry Study
Brief Title: INtravenous TNK for Acute isChemicsTroke in China
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Other Study IDs: y2020-022
Record Dates: First submitted 2020-10-03; First posted 2020-10-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: rhTNK-tPA — Thrombolysis

SUMMARY:
Acute ischemic stroke is the most common type of stroke, accounting for about 60%-80% of all stroke, with high incidence, high mortality, high disability rate, has become the first cause of death in China. At present, only ultra-early thrombolytic therapy, endovascular therapy and antiplatelet therapy have obtained evidence-based medical evidence in ischemic stroke treatment, but only thrombolytic therapy and endovascular therapy can improve the good prognosis of patients. Intravenous thrombolytic therapy within 4.5 hours after the onset of ischemic stroke symptoms has been shown to be effective, which is recommended in the guidelines.

In most countries, alteplase (R-tPA) is the only drug approved for the treatment of acute ischemic stroke. Recombinant human TNK tissue-type plasminogen activator (rhTNK-tPA) is a modified recombinant tissue-type plasminogen activator, with no procoagulant effect and a longer half life. In recent years, there are some studies on the comparison of therapeutic effects of TNK-tPA and RT-PA in patients with acute ischemic stroke, and TNK shows promising especially for large artery occlussion. At present, there are few reports on the application of rhTNK-tPA in Chinese stroke patients.

The aim of this study is to evaluate the efficacy and safety of rhTNK-tPA in Chinese patients with ischemic stroke in a prospective, multicenter registration study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 ;
2. The time from onset to treatment was less than 4.5 hours;
3. Ischemic stroke confirmed by head CT or MRI;
4. There are measurable neurological deficits;
5. First onset or previous onset without obvious sequelae (Mrs ≤1 score) ;
6. signed informed consent.

Exclusion Criteria:

1. Severe neurologic deficits before onset (mRS ≥2) ;
2. Significant head trauma or stroke in the last 3 months;
3. Subarachnoid hemorrhage;
4. A history of intracranial hemorrhage or head injury or acute stroke within 3 months;
5. Intracranial tumors, arteriovenous malformations or aneurysms;
6. Intracranial or spinal cord surgery within 3 months;
7. Non-compressible arterial puncture within 7 days;
8. Gastrointestinal or urinary tract hemorrhage within last 21 days;
9. Major surgery within 1 month;
10. Thrombocytopenia (platelet count <10×109/L);
11. Use of heparin or oral anticoagulation therapy within 48 hours;
12. Use of warfarin with an international normalised ratio >1.7 or PT >15 s;
13. Uncontrolled hypertension (SYSTOLIC >180 mmHg OR DIASTOLIC>110 mmHg) ;
14. The Blood Glucose concentration <50 mg/dl (2.7 mmol/L);
15. Severe systemic disease with poor life expectancy (<3 months); ;
16. Allergic to research drug;
17. Within 3 months or participating in other clinical trials;
18. Other conditions due to which investigators consider study participation inappropriate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute ischemic stroke patients who is eligible for intravenous thrombolysis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
The proportion of excellent prognosis (mRS 0-1) | 90 ± 7 days
  The proportion of excellent prognosis (mRS 0-1) after thrombolysis

SECONDARY OUTCOMES:
the proportion of good prognosis (mRS 0-2) | 90 ± 7 days
  The proportion of good prognosis (mRS 0-2) after thrombolysis
The incidence of stroke deterioration after thrombolysis | within 1 week
  NIHSS score increased by more than 2, excluding cerebral hemorrhage
the incidence of stroke recurrence and other vascular events | within 90 ± 7 days
  the incidence of stroke recurrence and other vascular events within 90 ± 7 days after thrombolysis
symptomatic intracerebral hemorrhage | within 36 hours
  any evidence of bleeding on the head CT scan associated with clinically significant neurological deterioration (NIHSS score ≥4 points increase)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China